CLINICAL TRIAL: NCT06204757
Title: Study of the Identification of Childbirth Trauma in the Birth Room by Midwives.
Acronym: TOPASE
Status: Active, not recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Other Study IDs: 2023/838
Record Dates: First submitted 2023-12-15; First posted 2024-01-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Trauma; Childbirth Problems
Keywords: trauma; delivery; childbirth; questionary
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- women: women who have given birth to a healthy baby
  Interventions: Other: questionary
- midwives
  Interventions: Other: questionary

INTERVENTIONS:
Other: questionary — questionary relating to birth trauma are completed by midwives and patients

SUMMARY:
Childbirth is a critical moment in this perinatal period, with high unpredictability and risks of medical complications for the mother and child. It can be experienced as a traumatic experience for the woman.

The consequences of a traumatic childbirth are numerous: psychiatric consequences for the mother: with increased risk of post-traumatic stress syndrome of postpartum depression decompensation of an old psychiatric illness, suicide , addictive disorders ; consequences on interactions: early mother-baby interactions are of poorer quality if the women have a negative experience of their birth.

Very few studies have focused on the early detection of traumatic childbirth, on the day of it. These evaluations only take into account the women's experience of their childbirth.

The systematization of a screening questionnaire for all deliveries would help to detect obvious traumatic deliveries but also to detect traumatic experiences when objectively the delivery occurs without obstetric complications.

This is why the objective of our study is to evaluate the perception of traumatic births by midwives.

DETAILED DESCRIPTION:
In a woman's life, the perinatal period is a phase of vulnerability, at risk of psychiatric complications: risk of decompensation of an existing psychiatric illness (depression, bipolar disorder, psychosis, anxiety disorder) and triggering of a pathology de novo. Childbirth is a critical moment in this perinatal period, with high unpredictability and risks of medical complications for the mother and child. It can be experienced as a traumatic experience for the woman. In France, 16.7% of women present major depressive symptoms 2 months after giving birth (National Institute of Health and Medical Research, 2021). Suicide is one of the two leading causes of maternal mortality up to 1 year postpartum, with approximately 1 suicide per month (approximately 13.4% of maternal deaths), the vast majority of which (91.3%) is considered potentially preventable (National Institute of Health and Medical Research, 2021b).

The data in the literature are still insufficient and lacking in homogeneity. Among the most relevant, an Australian study from 2014 found a traumatic childbirth experience in 14.3% of women (890 completed questionnaires) (Boorman et al., 2014). In recent studies, the rate of negative childbirth experiences ranges from 5 to 21% of women (Henriksen et al., 2017; Nystedt & Hildingsson, 2018; Sigurdardottir et al., 2017; Smarandache et al., 2016 ). The consequences of a traumatic childbirth are numerous:

* Psychiatric consequences for the mother: with increased risk of post-traumatic stress syndrome of postpartum depression decompensation of an old psychiatric illness, suicide (National Institute of Health and Medical Research, 2021a; Orsolini et al., 2016), addictive disorders.
* Consequences on interactions: early mother-baby interactions (first 4 months postpartum) are of poorer quality if the women have a negative experience of their birth.

Traumatic childbirth has long-term repercussions on identity, relationships with others, and adherence to care with more medical wandering.

It is therefore important to treat the trauma of childbirth early to reduce the severity and duration of its complications (Marianne Kédia & Sabouraud-Séguin, 2020).

If it is not identified in the maternity ward, women will often not talk about the trauma, or will talk about it after their next pregnancy. As mentioned above, the risk of depression and suicide is higher.

If it is identified on the day of the trauma, psychological or psychiatric support can be started during the stay in the maternity ward, by sharing this experience recognized by the healthcare teams. A single debriefing interview after a trauma is not enough to reduce the risk of complications but allows an alliance to be established to implement care (Sabouraud-Séguin, 2020).

The recognition of traumatic childbirth is recent, and teams are still insufficiently aware of the consequences, and poorly trained in the systematization of recommendations. Screening for traumatic childbirth should be carried out throughout the perinatal period. Before childbirth: during pregnancy monitoring, caregivers identify patients with vulnerabilities such as a history of trauma, complicated deliveries, or vulnerability. These women will be more at risk of having a negative experience of their childbirth (Ayers et al., 2016). In the delivery room: the teams identify obstetric situations at risk of trauma (instrument, cesarean section, somatic complications for the mother such as hemorrhages, and somatic complications for the child such as situations requiring neonatal resuscitation), and observe the reactions of the patient. During the stay in the maternity ward: the teams question the mothers' experience of childbirth, observe their behavior and first interactions. Symptoms that are part of the state of acute stress should alert you: intrusive symptoms, negative mood, dissociative symptoms, avoidance symptoms and arousal symptoms (American Psychiatric Association et al., 2015). After leaving the maternity ward, the woman has numerous follow-up appointments for herself and her baby, including the post-natal appointment. These moments of discussion are key moments for screening for traumatic symptoms (acute stress and post-traumatic stress syndrome) and depressive symptoms.

Very few studies have focused on the early detection of traumatic childbirth, on the day of it. These evaluations only take into account the women's experience of their childbirth. Two self-questionnaires were validated: Childbirth Experience Evaluation Questionnaire, QEVA (Carquillat et al., 2017; Chabbert et al., 2021); Peritraumatic Distress Inventory, PDI, which measures peri-traumatic distress, without being specific to an event, it is therefore not specialized for childbirth (Professional Space & Training | Info-Trauma, n.d.; Jehel et al., 2005 ).

The limits linked to self-questionnaires in a traumatic context and the impact of avoidance syndrome: women who have experienced a traumatic childbirth are more likely to avoid thinking about events, places, people linked to the trauma.

To our knowledge, no tool has been developed to assess the perception of traumatic births by midwives.

Midwives have an essential role during childbirth, from an obstetrical point of view, but also from a psychological point of view. They are present throughout the birth (labor, expulsion, delivery) and accompany the woman through her emotions, her doubts and her requests, with a common goal: the smooth running of the birth. However, they observe the entire course of the birth, with its complications and the reactions of the women. A hetero-assessment questionnaire, so that the trauma of childbirth can be assessed by midwives without needing the woman to recount her experience, would be useful for screening. The systematization of a screening questionnaire for all deliveries would help to detect obvious traumatic deliveries (for example during code red cesarean sections) but also to detect traumatic experiences when objectively the delivery occurs without obstetric complications.

In addition, the systematic questionnaire would make it possible to obtain the midwives' observations, which are not always transmitted in their entirety to the maternity team when the emotional experience has been too intense.

The objective of our study is to evaluate the perception of traumatic births by midwives.

The research hypothesis is that midwives can identify some indicators of birth trauma during childbirth and contribute to screening for traumatic birth.

ELIGIBILITY:
Inclusion Criteria:

* Women aged over 18
* Women followed after delivery in the maternity department of Besancon University Hospital
* Non-opposition indicating that the subject agrees to participate in the study and to comply with the requirements and restrictions inherent to this study
* Affiliation to a French social security scheme or beneficiary of such a scheme

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Subject unlikely to cooperate in the study and/or low cooperation anticipated by the investigator
* Language barrier preventing instructions from being understood
* Cognitive disorders preventing understanding of study instructions
* Subject without health insurance
* Women whose child is hospitalized in intensive care or has died

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: 1. women who gave birth to a healthy baby
  2. gynecological department midwife
Sampling Method: Probability Sample
Enrollment: 1440 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of midwives' perception of traumatic deliveries in relation to obstetrical data | within 12 hours of delivery.
  Using the Midwifery Trauma Assessment Questionnaire (QETRAS questionnaire) filled in by the midwife (who witnessed the child's expulsion) within 12 hours of delivery.

SECONDARY OUTCOMES:
Describe women's experiences of childbirth as measured by overall score on the QEVA self-questionnaire. | Between days 1 and 6 post-delivery
  Using Childbirth assessment self-questionnaire (QEVA self-questionnaire).
Describe women's experiences of childbirth as measured by Peri-traumatic distress inventory.Overall score on the PDI inventory | Between days 1 and 6 post-delivery
  Using Peri-traumatic distress inventory

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No